CLINICAL TRIAL: NCT00199602
Title: Prophylaxis of Thrombosis With Implantable Devices for Central Venous Access in Cancer Patients : Phase III Randomised Study
Brief Title: Prophylaxis of Thrombosis With Implantable Devices for Central Venous Access in Cancer Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: I99006
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2018-08-24 (Actual); Status verified 2008-12

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- lack of drug prophylaxis (No Intervention)
- HBPM 2500 UI anti Xa in one subcutaneous injection per day (Experimental)
  Interventions: Drug: warfarine - low molecular heparin
- warfarine 1mg daily (Experimental)
  Interventions: Drug: warfarine - low molecular heparin

INTERVENTIONS:
Drug: warfarine - low molecular heparin
  Arms: HBPM 2500 UI anti Xa in one subcutaneous injection per day; warfarine 1mg daily

SUMMARY:
This is a Phase III open-labed, multicenter, prospective, randomised study, and comparative 3-arms of 140 patients (i.e. 420 total patients).

Study period (date of first inclusion/last inclusion): 3 years Treatment period : 3 months

ELIGIBILITY:
Inclusion Criteria:

* First line chemotherapy for solid tumor with:
* Metastatic disease or
* Involved nodes or
* Unresectable tumor
* Indication for Implantable device for central venous access
* Potential survival > 3 months
* ECOG performance status 0 to 2 (WHO)
* Age between 18 and 75 years.
* Social security guaranteed
* Normal laboratory assessments (platelets> 100000/mm3, TP 60%, spontaneous TCA with M/T<1.5, TGO and TGP < 2xN, serum creatinin<120µmol/l)
* Informed consent signed

Exclusion Criteria:

* Inability to understand informed consent or interfering with compliance for treatment or protocol Anti-coagulant treatment -related criteria
* Acute infectious endocarditis
* History related with heparin allergy or thrombopenia due to heparin
* Uncontrolled high blood pressure (systolic blood pressure >180 mm Hg and/or diastolic blood pressure >110 mm Hg)
* Hemorrhagic syndrome ongoing
* Patient with platelet inhibitors treatment
* Chronic, daily treatment with anti-coagulant therapy (LMWH or AVK), use as preventive or curative level
* Patient with liver failure (TP<60%) or renal insufficiency (creatinin clearance< 20 ml/mn)
* Women with pregnancy and lactating Pathology-related criteria
* deep venous thrombosis history or pulmonary embolism (< 6 months)
* Clinical suspicious of brain metastasis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Actual)
Dates: Start 1999-08 (Actual); Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the prevalence of symptomatic or asymptomatic deep venous thrombosis in cancer patients with implantable device for central venous access with or without prophylaxis : | Day90
Low molecular weight Heparin (LMWH) 2500 U anti-XA/day or Warfarine 1 mg/day during the first line of chemotherapy | Day90

SECONDARY OUTCOMES:
- Detection of asymptomatic thrombosis related to implantable device estimated by a systematic echo-doppler. - | Day90
- Frequency of other symptomatic venous thromboembolic events between 3 groups. | J0, J1, J21, J42, J63 and J90
Comparison of thrombosis prophylaxis by LMWH with warfarin at low dose | Day90
-Costs in the 3 strategies | J90
- Tumoral response to chemotherapy in the 3 groups. | Day90
- Overall survival in each group. | Day90

CONTACTS AND LOCATIONS:
Overall Officials: Nicole TUBIANA-MATHIEU, MD, Principal Investigator — University Hospital, Limoges
Locations (1):
- Oncologie Médicale, Limoges, France

REFERENCES:
- [Result] Lavau-Denes S, Lacroix P, Maubon A, Preux PM, Genet D, Venat-Bouvet L, Labourey JL, Martin J, Slaouti P, Tubiana-Mathieu N. Prophylaxis of catheter-related deep vein thrombosis in cancer patients with low-dose warfarin, low molecular weight heparin, or control: a randomized, controlled, phase III study. Cancer Chemother Pharmacol. 2013 Jul;72(1):65-73. doi: 10.1007/s00280-013-2169-y. Epub 2013 May 1. PMID 23636449